CLINICAL TRIAL: NCT02990117
Title: An In-depth Understanding of Determinants of Inhaled ICS Treatment Compliance of Asthma Patients: Generate Data From Structured Patient Interview & Cross Sectional Survey
Brief Title: ICS Treatment Compliance of Asthma Patients
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Li Manxiang, Director, Respiratory department, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: ESR-16-12138
Record Dates: First submitted 2016-11-21; First posted 2016-12-13 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Asthma, Allergic
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Asthmatic patient: Asthma patients aged >18 in out-patient clinic of the first affiliated hospital of Xi'an Jiaotong university from November 2016 to January 2018 were investigated. A two-stage study was applied which was non-assumptive deep dive qualitative scoping to investigate the determinants of poor compliance in stage 1 asthma patients, and developed new questionnaire for cross sectional survey in stage 2 to obtain more accurate information about the critical issues on asthma management.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The introduction of inhaled medication as the primary treatment for asthma has led to substantial improvements in asthma control [1, 2]. However, uncontrolled asthma is still common and represents a considerable burden to patients and society [3, 4]. An important reason for poor asthma control and consequently, increased healthcare expenditure is suboptimal adherence to the prescribed regimen [5-7].

Real-world market research study in hospitals across China reported that physicians perceived that only 23% of patients were fully compliant with their medication regime (77% non-adherent), compared to 55% in the European Union and 63% in the US [AZ internal document]. The physician reported rate of full adherence was lower than the patient-reported rate (38%). Poor patient adherence was the challenge most frequently mentioned (by 41% of physicians) when treating an asthma.[8]

However

There is some evidence on the drivers of patient behaviour around low adherence but more depth research is needed

There is little evidence on variation of determinants of asthma inhaled treatment across different age of group

Our research aims to address above data gap Mean while this research can guide the development of new module on Red Scarf patient education program.

DETAILED DESCRIPTION:
Study site(s) and number of subjects planned 8 level-3 hospitals across West China will participate in this study. 40 not well controlled asthma patients will participate the structured interview in stage1 and a total number of 300 patients are expected to participate cross sectional survey in stage 2.

Study period Estimated Time CSP approved Oct. 2016 First subject in Jan. 2017 Last subject in Aug. 2017 Database lock Dec. 2017 CSR Mar. 2017

Study design It is study including 2 stage, stage 1 of structured patient interview by investigators, Stage 2 of a multi-center, cross-sectional survey. 40 eligible asthma patients and/or their family supporter will be invited to participate in a one-time face to face structured interview in stage 1. Around 350 eligible asthma patients will be invited to participate in cross sectional survey which all Information and relevant data of their compliance to inhaled treatment therapy and response to measurement of compliance risk factors (determinants explored from stage 1) will be collected according to CRF, and inputted into an on-line electronic questionnaire data capture (EDC) system by site investigator(s), and valid data will be taken into statistical analyses.

Target subject population Stage 1: Asthmatic patients with in adequate asthma control (defined by GINA partly or un-control due to inhaled treatment compliance (physician judgement) Stage 2: Asthmatic patient who visit the outpatient clinic will be interviewed by investigator.

Objectives

Stage 1:

Primary Objective: Outcome Measure:

Non- Assumptive Deep Dive Qualitative Scoping to investigate determinants of poor adherence to ICS treatment through structured interview & taskforce workshop Decide key measures for phase2 survey through steering committee group review. Categorized "risk factors" (patient behavior/belief, social status, medical care availability etc.) which very likely led to poor patient adherence on inhaled treatment adherence in partly or uncontrolled asthma patients

1. Therapy related factors
2. Patient related factors
3. Provider related factors
4. Disease related factors
5. Practice and system related factors

Questionnaire with measures for asthma patient adherence determinants in survey on stage 2

Stage 2:

Primary Objective: Outcome Measure:

To investigate the relationship different risk factors (determinants explored from stage 1) and treatment adherence to further identify top 5 determinants most closely relative to inhalation treatment adherence

Decide key measures for phase2 survey through steering committee group review. Asthma patient compliance level on Inhaled treatment (ICS or ICS/LABA) by using validated MARS-A scale questionnaire below.

Risk factors (determinants explored from stage 1) measurements response from asthma patients

Secondary Objective: Outcome Measure :

Similar objectives on deferent life-stage group of asthma patients. Similar analysis by different life-stage group of patients (18- 30, 31-45,45-60, 60+)

Statistical methods

* All results will be described. In general, the descriptive statistics (number, mean, and median, standard deviation, minimum and maximum) will be presented for continuous variables. The frequency and percentage of subjects at each level or category will be presented for categorical variables. Where appropriate, 95% confidence intervals will be constructed.
* Risk factor analysis will be performed using univariate and multivariate regression model to explore the relationship between risk factors and the compliance level. In addition to multivariate analysis using all variables, a step-wise variable selection can be used. The level of both variable inclusion and exclusion will be set as 0.15. The important variable (s) can be forced in the model if applicable.

ELIGIBILITY:
Inclusion Criterias:

1. Age ≥18 years old
2. Living in the city same as the study site for a minimum period of two years
3. Having China city residence medical insurance
4. A history of at least one year of diagnosed asthma who should be on ICS or ICS/LABA inhalation treatment based on the criteria established by GINA.
5. Patients On inhaled ICS or ICS/LABA treatment regard less of compliance level in the past 6 months
6. Subjects who are willing to sign the informed consent.

Exclusion Criteria:

1. Patients with active cardio or pulmonary disease such as bronchiectasis, COPD, cystic fibrosis, pulmonary tuberculosis, lung cancer, severe heart disease, etc.; other disorder such as HIV/AIDS, etc; or therapy that according to the physician could interfere with the aim of the study.
2. Patients with mental or neurological diseases, or due to alcohol or other drug abuse, that may be incapable to understand and answer the question honestly, or unwilling to do so.
3. Other conditions judged by investigator as unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 1: Asthmatic patients with in adequate asthma control (defined by GINA partly or un-control due to inhaled treatment compliance (physician judgement) Stage 2: Asthmatic patient who visit the outpatient clinic will be interviewed by investigator.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
MARS-A scale | Mar.2017-Dec,2017
  MARS-A scale is a valicated tool to assess inhaled treatment compliance of asthma patients Risk factors (determinants explored from stage 1) measurements response from asthma patients

SECONDARY OUTCOMES:
MARS-A scale of group patients age in 18- 30, age in 31-45, age in 45-60, age above 60 | Mar.2017-Dec,2017
  MARS-A scale is a valicated tool to assess inhaled treatment compliance of asthma patients Risk facto rs measurements response from asthma patients

CONTACTS AND LOCATIONS:
Overall Officials: Manxiang Li, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: Undecided